CLINICAL TRIAL: NCT02093156
Title: A Predictive Score Identifies Patients With Inadequate Bowel Preparation for Colonoscopy
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Other Study IDs: 20130910-3
Record Dates: First submitted 2014-03-19; First posted 2014-03-20 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Bowel Preparation; Ottawa Score
Keywords: bowel preparation; Ottawa Score

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- training cohort: the training cohort was used to establish the bowel preparation score (BPS)
  Interventions: Other: Bowel preparation instructions
- validation cohort: the validation cohort was used to verify the BPS (bowel preparation score)
  Interventions: Other: Bowel preparation instructions

INTERVENTIONS:
Other: Bowel preparation instructions — The same-day preparation method was used as previously reported. Briefly, all patients were instructed to have a regular diet for breakfast and lunch, but only clear liquids for dinner on the day before the colonoscopy. They were asked to drink two bags of PEG-ELP (polyethylene glycol electrolyte powder) dissolved in 2 L of water, or 45 mL of sodium phosphate be diluted in 240 mL of cool water follow with at least 1.5 L of water at 05:00-06:00 h within 2 h on the day of colonoscopy. Patients were encouraged to drink more clear liquids after purgatives for adequate hydration before colonoscopy.

SUMMARY:
Colonoscopy is the current standard method for evaluating the colorectal diseases. Adequate bowel preparation is essential for optimal visualization of the colorectal mucosa. However, inadequate bowel preparation (IBP) had been unexpectedly reported in up to 30% of patients undergoing colonoscopy. Many factors may influence the quality of bowel preparation, which can be broadly categorized as patient-related or procedure-related. It has been shown that split-dose regimen or some modified educational strategies can improve the quality of bowel preparation. For the patients with possible IBP before the performing of colonoscopy, it may be better to repeat bowel preparation with modified or enhanced strategies in case of failed intubation, missed lesions or unnecessarily increased cost. Thus, it is important to set up a model to predict the quality of bowel preparation individually.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-90 years old who undergoing colonoscopy

Exclusion Criteria:

* failed colonoscopy because of technical chanllenge or poor tolerance of patients
* history of colorectal surgery
* prior finding of severe colonic stricture or obstructing tumor
* dysphagia
* compromised swallowing reflex or mental status
* significant gastroparesis or gastric outlet obstruction or ileum
* known or suspected bowel obstruction or perforation
* pregnancy
* unable to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a prospective study involving two tertiary centers in China. The patients of the training cohort were enrolled from the Endoscopy Center of Xijing Hospital of Digestive Diseases in China. The patients of the validation cohort were enrolled from the Shaanxi Second People's Hospital in China.
Sampling Method: Non-Probability Sample
Enrollment: 605 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Adequate bowel preparation quality at the time of colonoscopy defined by Ottawa score<6 | up to 4 months
  Ottawa score：A)cleanliness of each part of the colon: 0=excellent 1=good 2=fair 3=poor 4=inadequate B)fluid in whole colon: small=0 moderate=1 large=2
  The bowel preparation was considered inadequate if (1) inadequate visualization on colonoscopy defined by Ottawa score≥6; (2) the colonoscopy was cancelled because of poor bowel preparation or personal reasons.

SECONDARY OUTCOMES:
Polyp detection rate | up to 4 months
  The proportion of participants with at least one polyp in each group

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Endoscopic center, Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi
  - Shaanxi Second People's Hospital, Xi'an, Shaanxi

REFERENCES:
- See also: Colonoscopy completion in a large safety net health care system — http://www.ncbi.nlm.nih.gov/pubmed/18304886
- See also: Bowel preparation with split-dose polyethylene glycol before colonoscopy: a meta-analysis of randomized controlled trials — http://www.ncbi.nlm.nih.gov/pubmed/21628016
- See also: Development and validation of a novel patient educational booklet to enhance colonoscopy preparation — http://www.ncbi.nlm.nih.gov/pubmed/?term=21483463
- See also: Telephone-based re-education on the day before colonoscopy improves the quality of bowel preparation and the polyp detection rate: a prospective, colonoscopist-blinded, randomised, controlled study — http://www.ncbi.nlm.nih.gov/pubmed/23503044
- See also: Impact of patient education with cartoon visual aids on the quality of bowel preparation for colonoscopy — http://www.ncbi.nlm.nih.gov/pubmed/22840295